CLINICAL TRIAL: NCT00006734
Title: Trial of Chemotherapy Intensification Through Compression in Ewing's Sarcoma and Related Tumors
Brief Title: Comparison of Combination Chemotherapy Regimens in Treating Patients With Ewing's Sarcoma or Neuroectodermal Tumor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEWS0031; COG-AEWS0031 (Other: Children's Oncology Group); CDR0000068323 (Other: Clinical Trials.gov); A7983 (Other: Children's Cancer Group)
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Sarcoma
Keywords: localized Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Doxorubicin; Etoposide; etoposide phosphate; Ifosfamide; Vincristine; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Brachytherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen A (Experimental): Test the hypothesis that chemotherapy given every two weeks (Regimen B) will produce higher event-free survival. Treatment will occur in two phases: Induction and Continuation, with 14 cycles of chemotherapy in all. Induction consists of the first twelve weeks (four cycles on Regimen A. The cycles alternate between vincristine sulfate, doxorubicin hydrochloride, cyclophosphamide, MESNA and ifosfamide, etoposide, MESNA. G-CSF (Filgrastim) is given between chemotherapy doses. Local control (Surgery, Radiation Therapy, or a combination) will begin on Week 13 which will be after four cycles of chemotherapy.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: vincristine sulfate; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: brachytherapy; Radiation: radiation therapy
- Regimen B (Experimental): Conventional every-three-week chemotherapy for patients with Ewing sarcoma and related tumors. Treatment will occur in two phases: Induction and Continuation, with 14 cycles of chemotherapy in all. Induction consists of the first twelve weeks six cycles on Regimen B). The cycles alternate between vincristine sulfate, doxorubicin hydrochloride, cyclophosphamide, MESNA and ifosfamide etoposide MESNA. G-CSF (Filgrastim) is given between chemotherapy doses. Local control (surgery, Radiation Therapy, or a combination) will begin on Week 13, which will be after six cycles of chemotherapy.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: vincristine sulfate; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: brachytherapy; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — Given IV
  Other Names: GRANULOCYTE COLONY-STIMULATING FACTOR; r-metHuG-CSF; G-CSF; Neupogen; NSC 614629
Drug: cyclophosphamide — Given IV
  Other Names: CTX; Cytoxan; NSC #026271
Drug: doxorubicin hydrochloride — Given IV
  Other Names: Adriamycin; NSC #123127; IND #7038
Drug: etoposide — Given IV
  Other Names: VP-16; VePesid; Etopophos; NSC #141540
Drug: ifosfamide — Given IV
  Other Names: Ifex; NSC #109724
Drug: vincristine sulfate — Given IV
  Other Names: Oncovin; NSC #067574
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which chemotherapy regimen combined with radiation therapy and/or surgery is more effective in treating Ewing's sarcoma or primitive neuroectodermal tumor.

PURPOSE: Randomized phase III trial to compare the effectiveness of different chemotherapy regimens combined with radiation therapy and/or surgery in treating patients who have Ewing's sarcoma or primitive neuroectodermal tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of interval-compressed vs standard chemotherapy in terms of event-free survival and overall survival in patients with newly diagnosed, localized Ewing's sarcoma or peripheral primitive neuroectodermal tumor.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (under 18 years vs 18 years and over) and location of primary disease (pelvic vs nonpelvic). Patients are randomized to 1 of 2 treatment arms for induction and continuation therapy.

* Induction therapy (weeks 1-12):

  * Arm I: Patients receive alternating courses of chemotherapy consisting of vincristine IV on day 1, doxorubicin IV continuously over 48 hours on days 1 and 2, and cyclophosphamide IV over 1 hour on day 1 for courses 1 and 3 and ifosfamide IV over 1 hour and etoposide IV over 1-2 hours on days 1-5 for courses 2 and 4. Beginning 24 hours after the last dose of chemotherapy for each course, patients receive filgrastim (G-CSF) subcutaneously (SC) daily until blood counts recover. Treatment continues every 3 weeks for 4 courses.
  * Arm II: Patients receive alternating courses of chemotherapy consisting of vincristine, doxorubicin, and cyclophosphamide as in arm I for courses 1, 3, and 5 and ifosfamide and etoposide as in arm I for courses 2, 4, and 6. Patients also receive G-CSF as in arm I. Treatment continues every 2 weeks for 6 courses.

After completion of induction therapy, patients in both arms receive local control treatment to the primary tumor. Patients receive continuation chemotherapy after surgery or concurrently with radiotherapy.

* Continuation therapy:

  * Arm I (weeks 13-42): Patients receive additional alternating courses of chemotherapy as in arm I of induction therapy with the exception of vincristine and cyclophosphamide alone for courses 7 and/or 11 and/or 13. Patients also receive G-CSF as in induction therapy. Treatment continues every 3 weeks for 10 courses.
  * Arm II (weeks 13-29): Patients receive additional alternating courses of chemotherapy as in arm II of induction therapy with the exception of vincristine and cyclophosphamide alone for courses 9 and/or 11 and/or 13. Patients also receive G-CSF as in induction therapy. Treatment continues every 2 weeks for 8 courses.

Patients are followed every 3 months for 4 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: Approximately 528 patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed localized Ewing's sarcoma or peripheral primitive neuroectodermal tumor (PNET) of the bone or soft tissues

  * Diagnostic biopsy of primary tumor within 30 days of study
* Paraspinal or bony skull tumors of extradural origin allowed

  * No intradural soft tissue tumors
* Askin's tumor of the chest wall allowed

  * Chest wall tumors with ipsilateral pleural effusions or ipsilateral pleural-based secondary tumor nodules allowed
  * No contralateral pleural effusions
* No metastatic disease or distant node involvement

  * One pulmonary or pleural nodule greater than 1 cm in diameter OR more than 1 nodule greater than 0.5 cm in diameter are considered pulmonary metastasis
  * Solitary lung nodules of 0.5-1 cm OR multiple nodules of 0.3-0.5 cm allowed unless biopsy positive for tumor
* Light microscopic appearance (hematoxylin and eosin stained) consistent with Ewing's sarcoma or peripheral PNET
* No immunohistochemical or ultrastructural evidence of rhabdomyosarcoma
* No esthesioneuroblastoma
* Clinically or pathologically involved regional lymph nodes allowed
* No CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 50 and under at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine normal for age
* Creatinine clearance or isotope glomerular filtration rate at least 75 mL/min

Cardiovascular:

* Shortening fraction at least 28% by echocardiography OR
* Ejection fraction at least 55% by radionuclide angiogram

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy except skin cancer diagnosed at least 5 years ago and currently in remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for skin cancer
* No concurrent sargramostim (GM-CSF)
* No concurrent pegfilgrastim

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* Prior complete or partial excision of primary tumor allowed

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 587 (Actual)
Dates: Start 2001-05; Primary Completion 2006-08 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Event-free survival | Time from study entry until disease progression, death without progression of disease, occurrence of a second malignant neoplasm or last follow-up, whichever comes first, assessed up to 5 years
  Assessed using a two sided log rank test of 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B. Womer, MD, Study Chair — Children's Hospital of Philadelphia
Locations (239):
- United States (212):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - General Robert Huyser Cancer Center at David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - St. Vincent Hospitals and Health Care Centers, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Pediatric Specialty Clinic at Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Walter Reed Army Medical Center, Silver Spring, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis/St. Paul, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - Children's Hospital of Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Valerie Fund Children's Center at Atlantic Health, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Children's Hospital at Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Comprehensive Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Dakota Cancer Institute at Innovis Health - Dakota Clinic, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Doernbecher Children's Hospital at Oregon Health & Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - Methodist Cancer Center at Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Cancer Care Center at Skagit Valley Hospital, Mount Vernon, Washington
  - Harborview Medical Center, Seattle, Washington
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Medical College of Ohio Cancer Institute, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- University Medical Center Groningen, Groningen, Netherlands
- Starship Children's Health, Auckland, New Zealand
- Puerto Rico (2):
  - Puerto Rico Cancer Center at University of Puerto Rico - Medical Sciences Campus, San Juan
  - San Jorge Children's Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Background] van Doorninck JA, Ji L, Schaub B, Shimada H, Wing MR, Krailo MD, Lessnick SL, Marina N, Triche TJ, Sposto R, Womer RB, Lawlor ER. Current treatment protocols have eliminated the prognostic advantage of type 1 fusions in Ewing sarcoma: a report from the Children's Oncology Group. J Clin Oncol. 2010 Apr 20;28(12):1989-94. doi: 10.1200/JCO.2009.24.5845. Epub 2010 Mar 22. PMID 20308669
- [Result] Womer RB, West DC, Krailo MD, Dickman PS, Pawel BR, Grier HE, Marcus K, Sailer S, Healey JH, Dormans JP, Weiss AR. Randomized controlled trial of interval-compressed chemotherapy for the treatment of localized Ewing sarcoma: a report from the Children's Oncology Group. J Clin Oncol. 2012 Nov 20;30(33):4148-54. doi: 10.1200/JCO.2011.41.5703. Epub 2012 Oct 22. PMID 23091096
- [Result] Borinstein SC, Barkauskas DA, Krailo M, Scher D, Scher L, Schlottmann S, Kallakury B, Dickman PS, Pawel BR, West DC, Womer RB, Toretsky JA. Investigation of the insulin-like growth factor-1 signaling pathway in localized Ewing sarcoma: a report from the Children's Oncology Group. Cancer. 2011 Nov 1;117(21):4966-76. doi: 10.1002/cncr.26112. Epub 2011 Apr 8. PMID 21480204
- [Result] Womer RB, West DC, Krailo MD, et al.: Randomized comparison of every-two-week v. every-three-week chemotherapy in Ewing sarcoma family tumors (ESFT). [Abstract] J Clin Oncol 26 (Suppl 15): A-10504, 2008.
- [Derived] Cash T, Krailo MD, Buxton AB, Pawel BR, Healey JH, Binitie O, Marcus KJ, Grier HE, Grohar PJ, Reed DR, Weiss AR, Gorlick R, Janeway KA, DuBois SG, Womer RB. Long-Term Outcomes in Patients With Localized Ewing Sarcoma Treated With Interval-Compressed Chemotherapy on Children's Oncology Group Study AEWS0031. J Clin Oncol. 2023 Oct 20;41(30):4724-4728. doi: 10.1200/JCO.23.00053. Epub 2023 Aug 31. PMID 37651654
- [Derived] Mora J, Castaneda A, Perez-Jaume S, Lopez-Pousa A, Maradiegue E, Valverde C, Martin-Broto J, Garcia Del Muro X, Cruz O, Cruz J, Martinez-Trufero J, Maurel J, Vaz MA, de Alava E, de Torres C. GEIS-21: a multicentric phase II study of intensive chemotherapy including gemcitabine and docetaxel for the treatment of Ewing sarcoma of children and adults: a report from the Spanish sarcoma group (GEIS). Br J Cancer. 2017 Sep 5;117(6):767-774. doi: 10.1038/bjc.2017.252. Epub 2017 Aug 8. PMID 28787430